CLINICAL TRIAL: NCT02575066
Title: Phase II Clinical Study of Concurrent Pazopanib for Non-metastatic Sarcoma Patients to be Treated With Radiotherapy, Localized in the Extremities, Trunk and Chest Wall or the Head and Neck Region (PASART-2)
Brief Title: Clinical Study of Concurrent Pazopanib and Radiotherapy for Non-metastatic Sarcoma Patients
Acronym: PASART-2
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: stopping rule
Sponsor: The Netherlands Cancer Institute (Other)
Collaborators: Royal Marsden NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M15PAS; DSSG02 (Other: Dutch Sarcoma Study Group)
Record Dates: First submitted 2015-09-16; First posted 2015-10-14 (Estimated); Last update posted 2019-06-27 (Actual); Status verified 2019-06

CONDITIONS: Sarcoma; Soft Tissue Sarcomas
Keywords: pazopanib; radiotherapy
MeSH Terms: conditions — Sarcoma | interventions — Radiotherapy; pazopanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- radiotherapy combined with pazopanib (Other): patients during the first part of the study received concurrent radiotherapy (25x2Gy) and pazopanib (QD 800 mg). The patients of the second part of the study will receive concurrent radiotherapy (18x2Gy) and pazopanib (QD 800 mg).
  Interventions: Radiation: external beam radiotherapy; Drug: pazopanib

INTERVENTIONS:
Radiation: external beam radiotherapy — external beam radiotherapy 25 x 2 Gy / 18 x 2 Gy
  Other Names: radiotherapy
Drug: pazopanib — pazopanib QD 800 mg

SUMMARY:
Radiotherapy (RT) alone is able to induce a clinically significant effect with a variable pathologic response (a pathological complete remission, pCR, defined as ≥ 95%, or ≤ 5% remaining visible tumour cells) in only about 10% of cases. A prior phase I study (PASART-1; NCT01985295) suggested that 25 x 2 Gy preoperative RT in combination with once daily 800mg oral pazopanib is feasible, while inducing tissue replacing tumor that can consist of fibrosis and necrosis in 40% of thus treated patients.

During this study, the interim analysis showed that the combination treatment of preoperative radiation with orally pazopanib is more effective than was anticipated. For this reason, the pazopanib dose of 800 mg once daily is maintained but the RT dose is reduced to 18x2Gy instead of 25x2Gy. Predominant aim of this RT dose reduction is lowering the wound complication risk after preoperative radiotherapy.

DETAILED DESCRIPTION:
Patients of the first part of the study received radiotherapy (25x2Gy) and pazopanib (QD 800 mg).

Patients of the second part of the study received/ will receive radiotherapy (18x2Gy) and pazopanib (QD 800 mg).

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed newly diagnosed intermediate to high grade soft tissue sarcoma localized to the extremities, trunk and chest wall or the head and neck area, for which the standard treatment is a combination of and radiotherapy and surgery(deep seated and/or > 5cm according to the RECIST 1.1 criteria and/or an anticipated close resection margin and/or grade II/III according to the WHO definition)
* Age ≥ 18 years
* WHO performance status of ≤ 1
* Able and willing to undergo blood sampling for PK and PD analysis
* Able to swallow and retain oral medication
* Able and willing to undergo MRI scanning
* Able and willing to undergo tumor biopsies
* Adequate organ functions as described by the laboratory findings in the table 1. For thyroid function, the T4 and TSH values must be within normal values of the range of the participating centers
* Written informed consent prior to performance of study-specific procedures or assessments and must be willing to comply with treatment and follow up.

Exclusion Criteria

* Prior malignancies; except another malignancy and disease-free for ≥ 5 years, or completely resected non-melanomatous skin carcinoma or successfully treated in situ carcinoma.
* Patients with recurrent sarcomas (even without prior radiotherapy)
* Ewing sarcoma and other PNET family tumors, rhabdomyosarcomas (both pediatric and adult), osteosarcomas
* Clinically significant gastrointestinal abnormalities which might interfere with oral dosing diagnosed
* Poorly controlled hypertension [defined as systolic blood pressure (SBP) of ≥140 mmHg or diastolic blood pressure (DBP) of ≥ 90mmHg]
* Unstable or serious concurrent condition (e.g., active infection requiring systemic therapy)
* Prolongation of corrected QT interval (QTc) > 480 msecs on ECG
* History of any of more of the following cardiovascular conditions within the past 6 months:
* Cardiac angioplasty or stenting
* Myocardial infarction
* Unstable angina
* Symptomatic peripheral vascular disease
* Coronary artery by-pass graft surgery
* Class II, III or IV congestive heart failure as defined by the New York Heart Association (NYHA)
* History of cerebrovascular accident, pulmonary embolism or untreated deep venous thrombosis (DVT) within the past 6 months
* Macroscopic hematuria
* Hemoptysis that is clinically relevant within 4 weeks of first dose of pazopanib
* Evidence of active bleeding or bleeding diathesis
* Prior major surgery or trauma within 28 days prior to first dose of study medication and/or presence of any non-healing wound, fracture, or ulcer
* Chemotherapy or radiation therapy within 2 weeks prior to the first dose of study medication
* Biological therapy or treatment with an investigational agent within 28 days or five half-lives, whichever is longer prior to the first dose of study medication
* Prohibited medications listed in the protocol for 14 days or five half-lives of a drug (whichever is longer) prior to visit 1 and for the duration of the study
* Known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to pazopanib
* Any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule; those conditions should be discussed with the patient before registration in the trial
* Female patients who are pregnant, breast-feeding or male or female patients of reproductive potential who are not employing an effective method of birth control

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2016-03-17 (Actual); Primary Completion 2019-03-20 (Actual); Study Completion 2019-03-20 (Actual)

PRIMARY OUTCOMES:
pathological near complete remission of the resected specimen which has been treated with radiotherapy | 6 weeks post treatment
  Proportion of patients with resection specimens demonstrating induction of a pathological (near) complete remission (≥ 95% tumor regression). Pathological (near) complete remission is defined as ≥ 95% replacement of tumor with other tissue, usually fibrosis and) in the resection specimen post combined pazopanib and radiotherapy treatment

SECONDARY OUTCOMES:
Incidence toxicities measured by NCI-CTCAE v4.0 (radiotherapy alone, pazopanib alone or both) measured from start of treatment until 6 weeks post-treatment | during treatment and up to 6 weeks post treatment
Rate of response as measured by RECIST v 1.1 at 4 weeks after completing radiotherapy | 4 weeks post treatment
Incidence of acute post-operative wound complications up to 3 weeks (+/- 1 week) after surgery as defined in section 6.1.3 and reference 29 (see also appendix XII) | up to 3 weeks post surgery

CONTACTS AND LOCATIONS:
Overall Officials: Rick Haas, MD, PhD, Principal Investigator — The Netherlands Cancer Institute
Locations (3):
- Netherlands (2):
  - Antoni van Leeuwenhoek, Amsterdam
  - Leids Universitair Medisch Centrum, Leiden
- Royal Marsden Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No